CLINICAL TRIAL: NCT03625050
Title: Efficacy and Safety of Chuna Manual Treatment as an Adjunctive Therapy After Total Knee Arthroplasty: A Study Protocol for a Single-Center, Randomized, Assessor Blind, Parallel-Group Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gachon University Gil Oriental Medical Hospital (Other)
Collaborators: Catholic Kwandong University (Other)
Responsible Party: Principal Investigator, Yun-Kyung Song, Sponsor-principle investigator, Gachon University Gil Oriental Medical Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISEE_2018_TKA_CN
Record Dates: First submitted 2018-07-31; First posted 2018-08-10 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Total Knee Replacement; Manipulation
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chuna + Usual care (Experimental)
  Interventions: Procedure: Chuna + Usual care(Celecoxib and esomeprazole)
- Usual care (Active Comparator)
  Interventions: Drug: Usual care(Celecoxib and esomeprazole)

INTERVENTIONS:
Procedure: Chuna + Usual care(Celecoxib and esomeprazole) — Chuna therapy (CT), 2 sessions/week, 4 weeks (8 sessions in total) Usual care therapy (UC, Celecoxib 200mg, qd and esomeprazole 20mg, qd), 4 weeks
  Usual care consists of physical therapy, CP based medications and patients education. Physical therapy consists of meridian muscle interferential current electricity (or meridian transcutaneous electricity) and hot pack (or infrared lamp).
  CT and UC group will receive the same UC regimen.
  Arms: Chuna + Usual care
Drug: Usual care(Celecoxib and esomeprazole) — Usual care therapy (UC, Celecoxib 200mg, qd and esomeprazole 20mg, qd), 4 weeks
  Usual care consists of physical therapy, CP based medications and patients education. Physical therapy consists of meridian muscle interferential current electricity (or meridian transcutaneous electricity) and hot pack (or infrared lamp).
  Arms: Usual care

SUMMARY:
Evaluate the efficacy and safety of Chuna treatment as an adjunctive therapy in patients with moderate pain following total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NRS of knee pain ≥4 during the 7 days after 3 months total knee replacement
* Patients who have agreed to trial participation and provided written informed consent

Exclusion Criteria:

* Those who have been diagnosed with certain serious diseases that can cause knee pain. : tumor, infectious or inflammatory disease, etc.
* Those taking analgesics for the purpose of relieving pain, fever and inflammation within 7 days
* Those with progressive neurological deficits or with severe neurological symptoms
* Those who have other chronic conditions that may interfere with the interpretation of treatment effects or outcomes : Cardiovascular disease, kidney disease, diabetic neuropathy, dementia, epilepsy, etc.
* Those who are not fit or unsafe to chuna therapy: clotting disorders, Those receiving anticoagulant therapy, Severe diabetes patients who are at risk of infection, severe cardiovascular disease
* Those who are participating in other clinical trials
* Those who have a history of participating in other clinical trials within one month
* Those who are difficult to write a research consent form
* Those who are judged to be inappropriate for the clinical study by the researchers.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline K-WOMAC score at week 4 | Week 0, Week 4
  Assess the recovery of knee function

SECONDARY OUTCOMES:
Change from baseline K-WOMAC score at every visit | Week 0, Week 2, Week 4, Week 8
  Assess the recovery of knee function
Change from baseline EQ-5D score at every visit | Week 0, Week 2, Week 4, Week 8
  EQ-5D is a tool developed for health-related quality of life (HRQoL) assessment, and is widely used in the health care sector. Scores range from -1, 'health worse than death' to 1, 'perfect health'. EQ-5D-5L has 5 dimensions covering current health status and functionality: mobility (M), self care (SC), usual activities (UA), pain/discomfort (PD), and anxiety/depression (AD), to be rated out of 5 grades (1, no problem; 2, slight problem; 3, some/moderate problem; 4, severe problem; 5, extreme problem).
Change from baseline Numeric rating scale score at every visit | Week 0, Week 2, Week 4, Week 8
  In pain measurement using NRS, patients are asked to rate their pain by selecting a number from 0 to 10 that best represents their pain severity between the anchors of 0 which indicates 'no pain', and 10 which indicates 'worst pain possible'.
Change from baseline in Physical Condition related with mobility at every visit | Week 0, Week 2, Week 4, Week 8, Week 12
  mobility (5 meters walking test at comfortable speed - 5mWT) (meters/second)
Change from baseline in Physical Condition related with endurance at every visit | Week 0, Week 2, Week 4, Week 8, Week 12
  endurance (Sit-to-stand test - STS) (seconds)
Change from baseline in Timed Up and Go Test at every visit | Week 0, Week 2, Week 4, Week 8, Week 12
  a functional test evaluating the time to rise from a chair, walk 3 meters, turn around, walk back to the chair and sit down (abnormal cut-off value >12 seconds).
Change from baseline in Alternative-Step Test at every visit | Week 0, Week 2, Week 4, Week 8, Week 12
  a functional test measuring clinical balance performance, and it has been shown to predict fall risk among elderly subjects (seconds)
Change from baseline in Range of motion score at every visit | Week 0, Week 2, Week 4, Week 8
  Compare flexion and extension angle using long arm goniometer between experimental and comparator group
Difference between the EuroQol Visual Analogue Scale (EQ-VAS) at each timepoint and baseline, respectively | Week 0, Week 2, Week 4, Week 8
  EQ-VAS uses a vertical 10cm line labeled at each end with scale anchors. EQ-VAS is used to indicate the patient's health state and patients are asked to mark a point that represents their health state between the anchors of 'worst health state' and 'best health state imaginable'. Scores are recorded in millimeters with a total range of 0-100 millimeters.
Cost per QALY(Quality Adjusted Life Years) gained | Week 0, Week 4, Week 8, Week 12
  The quality of life estimation for QALY calculation will use the quality of life derived from EQ-5D as the main evaluation variable, and the calculation method is using Area under the curve method

CONTACTS AND LOCATIONS:
Overall Officials: Yun Kyung Song, PhD, Principal Investigator — Gachon university of Gil oriental hospital
Locations (1):
- Catholic Kwandong University International St. Mary'S Hospita, Incheon, South Korea